CLINICAL TRIAL: NCT00868478
Title: Phase I-II Trial of the Anti CD74 Monoclonal Antibody-Milatuzumab as a Single Agent in Refractory Chronic Lymphocytic Leukemia
Brief Title: The Humanized Monoclonal Antibody Milatuzumab for Refractory Chronic Lymphocytic Leukemia (CLL)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Dr. Michal Haran, Kaplan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMC-07-0080-CTIL
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: humanized monoclonal antibody
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — milatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Milatuzumab — Milatuzumab will be given at a starting dose of 120 mg/m2, and then if no response or significant toxicity is seen after a total of 12 weeks, the dose will be gradually increased, by 120 mg/ m2 every four weeks, for a total of another 12 weeks.
  Other Names: hLL1

SUMMARY:
The purpose of this study is to determine whether Milatuzumab is effective in patients with refractory chronic lymphocytic leukemia, and also to find out in which range of doses is a response seen.

DETAILED DESCRIPTION:
The aim of this study is to determine whether the anti-CD74 monoclonal antibody Milatuzumab provides benefit to subjects with CLL in advanced stage or progressive disease. The primary objectives of this study are to assess response rate to the agent, as well as the safety in CLL, using different doses: Overall response (OR), complete response (CR) and partial response (PR) will be determinate according to the NCI criteria.

The secondary objectives are to determine: duration of response, time to progression, overall survival, and the range of doses in which efficacy is seen and MTD not reached.

This study will be done in parallel with other phase I-II studies conducted by Immunomedics.

The study design will take into account that the high levels of circulating CD74expressing cells in CLL may affect both the acute (although probably not long term) toxicity and the efficacy of the study medication. This could translate to a different MTD and a different cumulative dose of Milatuzumab, needed to achieve response.(either a higher dose or longer treatment period.).

The study will be divided into two treatment phases. In the first phase we aim to address whether the dose of 120 mg/m2 is effective in CLL, and also if it is safe. In the second phase we will assess the safety and possible efficacy of higher doses, in those patients that did not achieve a significant response in the first phase. This will be done by gradual dose escalations, not to exceed 600 mg, or the MTD reached in other studies.

In addition, the study will aim at gaining further understanding of the effect of Milatuzumab on the biological in-vitro function of CLL cells.

ELIGIBILITY:
Inclusion Criteria:

* B-CLL confirmed according to NCI criteria
* CLL relapsed or refractory to prior antineoplastic therapy
* Signs of progressive disease; at least one:

  * B symptoms
  * lymphocyte doubling time of < 6 months
  * symptomatic lymphadenopathy or splenomegaly
  * cytopenias due to bone marrow failure)
* Age > 18 years, and less then 80
* Serum ALAT, ASAT, bilirubin, creatinine < 2x upper limit of normal
* Life expectancy > 6 months
* Patient's written informed consent

Exclusion Criteria:

* Active bacterial or viral infection
* Hypersensitivity to humanized monoclonal antibodies
* Concurrent antineoplastic treatment for CLL or other malignant disease
* Absolute neutrophil count < 1.5 K/

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Response to treatment | 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michal Haran, MD, Principal Investigator — Kaplan Medical Center
Locations (1):
- Kaplan Medical Center, Rehovot, Israel

REFERENCES:
- [Background] Binsky I, Haran M, Starlets D, Gore Y, Lantner F, Harpaz N, Leng L, Goldenberg DM, Shvidel L, Berrebi A, Bucala R, Shachar I. IL-8 secreted in a macrophage migration-inhibitory factor- and CD74-dependent manner regulates B cell chronic lymphocytic leukemia survival. Proc Natl Acad Sci U S A. 2007 Aug 14;104(33):13408-13. doi: 10.1073/pnas.0701553104. Epub 2007 Aug 8. PMID 17686984